CLINICAL TRIAL: NCT01424319
Title: Reducing Residual Albuminuria in Subjects With Diabetes & Nephropathy With Atrasentan - A Phase 2b, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Safety & Efficacy in Japanese Subjects
Brief Title: Reducing Residual Albuminuria in Subjects With Diabetes and Nephropathy With Atrasentan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-812
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease; Diabetic Nephropathy
Keywords: Endothelin Receptor Antagonists; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Proteinuria | interventions — Atrasentan; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-627, Low dose (Experimental)
  Interventions: Drug: Atrasentan low dose group
- ABT-627, High dose (Experimental)
  Interventions: Drug: Atrasentan high dose group
- ABT-627, Placebo (Placebo Comparator)
  Interventions: Drug: Atrasentan placebo group

INTERVENTIONS:
Drug: Atrasentan low dose group — Subjects will take two tablets daily of one of those which are atrasentan low dose, atrasentan high dose or atrasentan placebo for 12 weeks during the treatment period.
  Arms: ABT-627, Low dose
Drug: Atrasentan high dose group — Subjects will take two tablets daily of one of those which are atrasentan low dose, atrasentan high dose or atrasentan placebo for 12 weeks during the treatment period.
  Arms: ABT-627, High dose
Drug: Atrasentan placebo group — Subjects will take two tablets daily of one of those which are atrasentan low dose, atrasentan high dose or atrasentan placebo for 12 weeks during the treatment period.
  Arms: ABT-627, Placebo

SUMMARY:
Prospective, randomized, double-blind, placebo controlled, 12-week, multicenter study. The objective of the study is to evaluate the efficacy and safety of once daily administration of atrasentan tablets compared to placebo in reducing residual albuminuria in Japanese Type 2 diabetic patients with nephropathy who are treated with the maximum tolerated labeled dose for hypertension of a RAS (renin angiotensin system) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Type 2 diabetes and has been treated with at least one anti-hyperglycemic medication within the 12 months prior to the screening period.
* Patient is receiving a maximum tolerated labeled dose of an ACEi (Angiotensin Converting Enzyme inhibitor) or ARB (Angiotensin II Receptor Blocker)(Renin Angiotensin System (RAS) inhibitor). Estimated GFR (Glomerular Filtration Rate) is greater than or equal to 30 and less than or equal to 75 mL/min/1.73m2 by the CKD (chronic kidney disease)
* Epidemiology Collaboration (EPI) formula.
* UACR (Urinary Albumin to Creatinine Ratio) is greater than or equal to 200 mg/g as determined by the geometric mean of the three morning void urine specimens obtained at Run-in period.
* Serum albumin is greater than or equal to 3.0 g/dL. BNP (B-type Natriuretic Peptide) is less than or equal to 200 pg/mL.
* SBP (Systolic Blood Pressure) is greater than or equal to 110 mmHg and less than or equal to 160 mmHg. HbA1c (Glucosylated Hemoglobin A1c) is less than or equal to 12% and serum potassium is less than or equal to 5.5 mEq/L.

Exclusion Criteria:

* Patient has a history of moderate or severe edema, facial edema unrelated to trauma, or a history of myxedema in the prior 6 months to screening.
* Patient is receiving loop diuretics greater than or equal to 120 mg QD (Once Daily) of furosemide or greater than or equal to 3.0 mg QD (Once Daily) of bumetanide or greater than or equal to 150 mg QD (Once Daily) of ethacrynic acid or greater than or equal to 60 mg QD (Once Daily) of torasemide.
* Patient has a documented history of Stage C or Stage D heart failure, defined ACC/AHA (American College of Cardiology/ American Heart Association Practice Guidelines).
* Patient is receiving any of a combination of an ACEi (Angiotensin Converting Enzyme inhibitor) and ARB (Angiotensin II Receptor Blocker) or rosiglitazone or aliskiren or an aldosterone antagonist and patient is receiving pioglitazone and edema is present.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The change from baseline to each post-baseline visit in log-transformed UACR (urinary albumin to creatinine ratio) | Up to Week 12

SECONDARY OUTCOMES:
The proportion of subjects who have achieved at least 30% reduction on UACR (Urinary Albumin to Creatinine Ratio) who have not had any form of treatment-emergent edema with moderate or severe severity. | Up to Week 12
The change from baseline to each post-baseline visit on log-transformed UACR (Urinary Albumin to Creatinine Ratio) and estimated GFR (Glomerular Filtration Rate) | Up to Week 12
The proportion of subjects who achieve various percent of reduction in UACR (Urinary Albumin to Creatinine Ratio) from baseline to final | Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Mosleh UDDIN, PharmD, Study Director — Abbott Japan Co.,Ltd
Locations (18):
- Japan (18):
  - Site Reference ID/Investigator# 62022, Azumino
  - Site Reference ID/Investigator# 58124, Chiba
  - Site Reference ID/Investigator# 57486, Fujisawa
  - Site Reference ID/Investigator# 55097, Ibaraki
  - Site Reference ID/Investigator# 56982, Ina
  - Site Reference ID/Investigator# 55093, Kawagoe
  - Site Reference ID/Investigator# 57485, Kawasaki
  - Site Reference ID/Investigator# 55092, Kōriyama
  - Site Reference ID/Investigator# 56524, Matsumoto
  - Site Reference ID/Investigator# 57242, Nagano
  - Site Reference ID/Investigator# 55781, Nagoya
  - Site Reference ID/Investigator# 60965, Nagoya
  - Site Reference ID/Investigator# 55304, Suwa
  - Site Reference ID/Investigator# 59474, Tokyo
  - Site Reference ID/Investigator# 59967, Ueda
  - Site Reference ID/Investigator# 55095, Yokohama
  - Site Reference ID/Investigator# 57484, Yokohama
  - Site Reference ID/Investigator# 59842, Yokohama

REFERENCES:
- [Result] de Zeeuw D, Coll B, Andress D, Brennan JJ, Tang H, Houser M, Correa-Rotter R, Kohan D, Lambers Heerspink HJ, Makino H, Perkovic V, Pritchett Y, Remuzzi G, Tobe SW, Toto R, Viberti G, Parving HH. The endothelin antagonist atrasentan lowers residual albuminuria in patients with type 2 diabetic nephropathy. J Am Soc Nephrol. 2014 May;25(5):1083-93. doi: 10.1681/ASN.2013080830. Epub 2014 Apr 10. PMID 24722445
- [Result] Kohan DE, Lambers Heerspink HJ, Coll B, Andress D, Brennan JJ, Kitzman DW, Correa-Rotter R, Makino H, Perkovic V, Hou FF, Remuzzi G, Tobe SW, Toto R, Parving HH, de Zeeuw D. Predictors of Atrasentan-Associated Fluid Retention and Change in Albuminuria in Patients with Diabetic Nephropathy. Clin J Am Soc Nephrol. 2015 Sep 4;10(9):1568-74. doi: 10.2215/CJN.00570115. Epub 2015 Jul 7. PMID 26153128
- [Derived] Lin CW, Mostafa NM, L Andress D, J Brennan J, Klein CE, Awni WM. Relationship Between Atrasentan Concentrations and Urinary Albumin to Creatinine Ratio in Western and Japanese Patients With Diabetic Nephropathy. Clin Ther. 2018 Feb;40(2):242-251. doi: 10.1016/j.clinthera.2017.07.011. Epub 2017 Jul 27. PMID 28756065